CLINICAL TRIAL: NCT05828745
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Ascending Doses of CB06-036 in Subjects With Chronic Hepatitis B
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CB06-036 in Subjects With Chronic Hepatitis B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Zhimeng Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CB06-036-102
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-08

CONDITIONS: Chronic Hepatitis b
Keywords: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- CB06-036 Cohort 1 (Experimental): CB06-036 1.5 mg once weekly
  Interventions: Drug: CB06-036
- Placebo Cohort 1 (Placebo Comparator): Placebo 1.5 mg once weeky
  Interventions: Drug: Placebo
- CB06-036 Cohort 2 (Experimental): CB06-036 3.0 mg once weekly
  Interventions: Drug: CB06-036
- Placebo Cohort 2 (Placebo Comparator): Placebo 3.0 mg once weekly
  Interventions: Drug: Placebo
- CB06-036 Cohort 3 (Experimental): CB06-036 1.5 mg twice-a-week, for 4 weeks
  Interventions: Drug: CB06-036
- Placebo Cohort 3 (Placebo Comparator): Placebo 3.0 mg twice-a-week, for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CB06-036 — CB06-036 capsule
  Arms: CB06-036 Cohort 1; CB06-036 Cohort 2; CB06-036 Cohort 3
Drug: Placebo — Placebo capsule
  Arms: Placebo Cohort 1; Placebo Cohort 2; Placebo Cohort 3

SUMMARY:
CB06-036 is an investigational drug developed by Shanghai Zhimeng Biopharma Inc. for the treatment of Chronic Hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provide written informed consent before any study assessment is performed. 2. Male or nonpregnant, nonlactating female between the ages of 18 and 65 years (inclusive) at screening.

Females of childbearing potential (as defined in Appendix 3) must have a negative serum pregnancy test at screening and a negative urine or serum pregnancy test at baseline prior to enrollment and agree to use 2 methods of birth control. Methods must include 1 highly effective method with a secondary method of birth control during the study and for 3 months following the last dose of CB06-036. These methods are defined in Appendix 3.

Note: Females must agree not to breastfeed during the study and 30 days after receiving the last administration of CB06-036 and not to donate eggs (ova, oocytes) for assisted reproduction during the study and 90 days after receiving the last administration of CB06-036. Females of nonchildbearing potential defined as permanently sterile (ie, due to hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or postmenopausal, as defined in Appendix 3.

Males with a female partner(s) of childbearing potential will agree to use contraception as detailed in Appendix 3. Male subjects must not donate sperm during the study and for at least 90 days after the last administration of CB06-036.

3. Documented evidence of chronic HBV infection (eg, HBsAg positive for more than 6 months) with detectable HBsAg level at screening. Cohort 4 only: qHBsAg should be <3000 IU/mL.

4. Have been on commercially available HBV NA treatment(s) (tenofovir alafenamide, tenofovir disoproxil fumarate, entecavir, either as a single agent or in combination) for at least 6 months with no change in regimen for 3 months prior to screening.

5. HBV DNA <90 IU/mL; measured at least once by local laboratory assessment within 6 months prior to screening.

6. HBV DNA <90 IU/mL at screening. 7. Body mass index (BMI) of 18.0 to 32.0 kg/m2 (inclusive), and a total body weight ≥50.0 kg for males and ≥45.0 kg for females at screening.

8. Electrocardiogram (ECG) without clinically significant abnormalities and with QT interval corrected using Fridericia's formula (QTcF) ≤450 msec for males and ≤470 msec for females at screening.

9. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures as specified in the protocol.

Exclusion Criteria:

* 1. CHB patients with extensive bridging fibrosis or cirrhosis (METAVIR ≥3 or Ishak ≥4 by a liver biopsy within 5 years, FibroTest score >0.48 and APRI >1, or a historic FibroScan >9 kPa within 6 months prior to screening).

  2. Subjects met any of the following laboratory parameters at screening:
  1. hemoglobin <12 g/dL (for males) or <11 g/dL (for females)
  2. white blood cell count <2500 cells/mm3 Protocol CONFIDENTIAL Labcorp Drug Development Study: 000000244098 Protocol Reference: CB06-036-102 Protocol Version 1.0, 24 January 2023 Page 8 of 68
  3. neutrophil count <1500 cells/mm3 (or <1000 cells/mm3 if considered a physiological variant in a subject of African descent)
  4. ALT >2 × ULN
  5. INR >ULN unless the subject is stable on an anticoagulant regimen affecting INR
  6. albumin <3.5 g/dL
  7. direct bilirubin >1.5 × ULN
  8. platelet Count <100,000/μL
  9. estimated creatinine clearance (CrCl) <60 mL/min (using the Cockcroft-Gault method).

     3.Active systemic infections (other than common cold) within 2 weeks before randomization.

     4.At screening, known history of lymphoma, leukemia, or malignancy within the past 5 years, except for squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.

     5.History or suspicion of hepatocellular carcinoma (ie, elevated alpha fetoprotein (AFP) >50 ng/mL; suggestive lesions on abdominal ultrasound or other imaging).

     6.History or presence of a medical condition associated with liver disease other than HBV infection (eg, hemochromatosis, autoimmune hepatitis, alcoholic liver disease, toxin exposure, thalassemia, moderate to severe nonalcoholic steatohepatitis). Other known clinically significant hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).

     7.History of transaminase (ALT and/or AST) flare in the previous 6 months prior to study enrollment.

     8.Personal or familial history or symptomatology indicative of a risk of immune mediated disease (eg, inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis, autoimmune uveitis, multiple sclerosis).

     9.Received a solid organ or bone marrow transplant. 10.Received prolonged systemic therapy with immunomodulators (eg, corticosteroids) or biologics (eg, monoclonal antibody, interferon) within 3 months of screening.

     11.Blood donation of approximately 500 mL within 56 days prior to first administration of study drug, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening.

     12.Have a known history of asthma. Note: Subjects with resolved childhood asthma with no history of hospitalization due to asthma are allowed.

     13.Current use of strong and moderate CYP3A4 inhibitors or inducers; please see Appendix 6 for a list.

     14.Are currently enrolled in, or discontinued from, a clinical trial involving an investigational product or non-approved drug within the last 4 weeks or at least 5 half-lives of the last dosing, if the half-life of the investigational product or non-approved drug is greater than 5 days; or concurrently enrolled in any other types of medical research judged not to be scientifically or medically compatible with this study.

     15.live vaccination during the course of the study, or have participated in a vaccine clinical trial within 12 weeks prior to randomization. Investigators should review the vaccination status of the subjects and follow the local guidelines for adult vaccination with non-live vaccines intended to prevent infectious disease prior to administration of study drug.

     16.Co-infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis D virus (HDV).

     • Subjects who are HCV Ab positive, but have a documented negative HCV RNA, are eligible.

     17.Abnormal clinical laboratory values at screening that, in the opinion of the investigator, pose an unacceptable risk to the subject or of interfering with the interpretation of study results if participating in the study.

     18.Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin laboratory test at screening or at Days -7 to -4.

     19.Have any other condition that precludes the subject from following and completing the protocol in the opinion of the investigator.

     20.Significant history or clinical manifestation of any metabolic, allergic, dermatologic, hepatic, renal, hematologic, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, retinal, or psychiatric disorder, as determined by the investigator (or designee).

     21.History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).

     22.Use or intend to use any nonprescription medications or products including vitamins, minerals, and herbal supplements (ie, traditional Chinese medicine), protein powders or fish oils preparations within 7 days prior to screening, considered to potentially impact subject safety or the objectives of the study, as determined by the investigator (or designee).

     23.Alcohol consumption of >21 units per week for males and >14 units for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.

     24.Ingestion of Seville orange or grapefruit-containing foods or beverages within 7 days prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of CB06-036 following multiple oral dose administration of CB06-036 in virally suppressed subjects with CHB. | From the date the first subject signs an informed consent form to the date of the last subject's last assessment (scheduled or unscheduled).
  Number of participants with treatment-related adverse events as assessed by CTCAE V5.0 or higher

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of CB06-036 following multiple oral dose administration in virally suppressed subjects with CHB. | From 30 minutes pre-dose to 24 hours post-dose
  Plasma will be collected at multiple timepoints from within 30 minutes pre-dose to 24 hours post-dose
Area Under the Plasma Concentration Versus Time Curve (AUC) of CB06-036 | From 30 minutes pre-dose to 24 hours post-dose
  Cohort1 & Cohort2: Plasma will be collected on Day 1 and Day 22 at multiple timepoints from within 30 minutes pre-dose to 24 hours post-dose.
  Cohort 3: Plasma will be collected on Day 1 and Day 25 at multiple timepoints from within 30 minutes pre-dose to 24 hours post-dose.
The following inflammatory cytokines and chemokines will be analyzed in serum: CCL11 (Eotaxin-1), CCL2 (MCP1), CCL20 (MIP3α), CCL4 (MIP1ß), CCL8 (MCP2), CRP, CXCL10 (IP10), CXCL8 (IL-8), CXCL9 (MIG), IFN-γ, IL-12p40, IL-12p70, IL-1RA, SAA, TNF-α | From pre-dose to 72 hours post-dose of the last dose of study drug
  Cohort1 & Cohort2: Blood samples will be collected on Day 1 and Day 22 at pre-dose and 2, 4, 8, 12, 48, and 72 hours post-dose.
  Cohort3: Blood samples for the PD of CB06-036 will be collected on Day 1 and Day 25 at pre-dose and 2, 4, 8, 12, and 48 hours post-dose. Also, the samples will be collected at Day 4 at pre-dose and 4 hours (peak) post-dose.

CONTACTS AND LOCATIONS:
Locations (2):
- First Hospital of Jilin University, Changchun, Jilin, China
- PCRN Trials Limited, trading as PCRN Auckland, Level 2, 2 Fred Thomas Drive, Takapuna, Auckland, 0622, New Zealand (hereinafter referred to as "Institution"), Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No